CLINICAL TRIAL: NCT00651599
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study Investigating the Efficacy and Tolerability of Angeliq(drospirenon2mg and Estradiol 1mg) in Postmenopausal Korean Women With Vasomotor Symptoms Over 3, 28 Day Treatment Cycle
Brief Title: Treatment of Vasomotor Symptoms in Korean Post Menopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91354; 308381
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Vasomotor Symptoms
Keywords: Vasomotor symptoms; Vasomotor System
MeSH Terms: interventions — estradiol-drospirenone combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 1 (Experimental)
  Interventions: Drug: Angeliq (Drospirenone/17ß-estradiol, BAY86-4891)

INTERVENTIONS:
Drug: Angeliq (Drospirenone/17ß-estradiol, BAY86-4891) — Treatments will be administered daily, orally during the whole treatment period of 16 weeks without a treatment-free interval.
  Arms: Arm 1
Drug: Placebo — Placebo treatments will be administered daily, orally during the whole treatment period of 16 weeks without a treatment-free interval.
  Arms: Arm 2

SUMMARY:
Study to demonstrate that the therapeutic efficacy of Angeliq® is better than placebo in Korean postmenopausal women with hot flushes and other climacteric symptoms. Safety and tolerability of Angeliq.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Korean women suffering from hot flushes

Exclusion Criteria:

* Standard exclusion criteria for HRT clinical trials had to be obeyed, including current or history of hormone dependent malignant disease, thromboembolic disorders, abnormal cervical smear, undiagnosed vaginal bleeding.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-07; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Hot flush (frequency and severity) | Daily in pre-treatment and treatment period

SECONDARY OUTCOMES:
Menopausal symptoms | Baseline and after 4 weeks, 8, 12 and 16 weeks of treatment
Urogenital symptoms | Baseline and after 4 weeks, 8, 12 and 16 weeks of treatment
Assessment of bleeding | daily in pre-treatment and treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Seoul, South Korea